CLINICAL TRIAL: NCT04209543
Title: A Randomized Double-blind Placebo Controlled Phase 3 Trial to Evaluate the Efficacy and Safety of Estetrol for the Treatment of Moderate to Severe Vasomotor Symptoms in Postmenopausal Women (E4Comfort Study I)
Brief Title: Estetrol for the Treatment of Moderate to Severe Vasomotor Symptoms in Postmenopausal Women (E4Comfort Study I)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Estetra (Industry)
Collaborators: ICON Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MIT-Do001-C301
Record Dates: First submitted 2019-12-20; First posted 2019-12-24 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-10

CONDITIONS: Vasomotor Symptoms; Menopausal Symptoms
Keywords: Estetrol; Hot Flushes; Vasomotor Symptoms
MeSH Terms: conditions — Hot Flashes | interventions — Estetrol; Progesterone

STUDY DESIGN:
Intervention Model Description: This study consists of 3 blinded arms (efficacy part) and 1 open-label arm (safety part).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study consists of 3 blinded arms (efficacy part) and 1 open-label arm (safety part).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Estetrol 15 mg - Efficacy Part (Experimental): Estetrol (E4) 15 mg was administered orally once daily for a minimum of 12 weeks and not longer than 13 weeks.
  Interventions: Drug: Estetrol
- Estetrol 20 mg - Efficacy Part (Experimental): Estetrol (E4) 20 mg was administered orally once daily for a minimum of 12 weeks and not longer than 13 weeks.
  Interventions: Drug: Estetrol
- Placebo - Efficacy Part (Placebo Comparator): Placebo was administered orally once daily for a minimum of 12 weeks and not longer than 13 weeks.
  Interventions: Drug: Placebo
- Estetrol 20 mg + P4 100 mg - Safety Part (Experimental): Estetrol (E4) 20 mg and Progesterone (P4) 100 mg was administered once daily for up to 53 weeks.
  Interventions: Drug: Estetrol; Drug: Progesterone

INTERVENTIONS:
Drug: Estetrol — Estetrol oral tablet: administered orally once daily
  Arms: Estetrol 15 mg - Efficacy Part; Estetrol 20 mg + P4 100 mg - Safety Part; Estetrol 20 mg - Efficacy Part
Drug: Placebo — Placebo oral tablet: administered orally once daily
  Arms: Placebo - Efficacy Part
Drug: Progesterone — Progesterone oral tablet: administered orally once daily
  Arms: Estetrol 20 mg + P4 100 mg - Safety Part

SUMMARY:
This is a two-part study designed to evaluate the effect of Estetrol (E4) 15 or 20 mg, or placebo on the severity and frequency of vasomotor symptoms (VMS) (Efficacy Study Part) and the safety of E4 20 mg (Endometrial and General Safety Study Part)

DETAILED DESCRIPTION:
This study consists of two-parts, performed with 2 separate groups of participants:

• Efficacy Study Part: Designed to evaluate the frequency and severity of vasomotor symptoms [VMS] in both hysterectomized and non-hysterectomized postmenopausal participants after treatment with E4 15 mg or 20 mg or placebo for up to 13 consecutive weeks. For endometrial protection, all non-hysterectomized participants were treated with 200 mg progesterone (P4) once daily for 14 consecutive days, after completion of the E4/placebo treatment. This part of the study consisted of 3 treatment groups.

• Safety Study Part: The Endometrial and General Safety Study Part is designed to evaluate the general safety, endometrial safety, secondary efficacy (lipid, glucose metabolism, health-related quality of life (HRQoL) and treatment satisfaction) of E4 in non-hysterectomized participants. All participants received E4 20 mg in combination with 100 mg P4 continuously for up to 53 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent form and any required privacy authorization prior to the initiation of any trial procedure, after the nature of the trial has been explained according to local regulatory requirements;
* Females, ≥ 40 up to ≤ 65 years of age at randomization;
* For hysterectomized subjects: documented hysterectomy must have occurred at least 6 weeks prior to the start of screening. Hysterectomy can be total or subtotal (i.e., cervix was not removed);
* For non-hysterectomized subjects: uterus with bi-layer endometrial thickness ≤ 4 mm on TVUS;
* For non-hysterectomized subjects: an evaluable endometrial biopsy taken during screening that reveals no abnormal results, i.e., presence of hyperplasia (simple or complex, with or without atypia), presence of carcinoma, and presence of disordered proliferative endometrium findings. The screening biopsy should have sufficient endometrial tissue for diagnosis;
* Seeking treatment for relief of VMS associated with menopause;

  1. For the Efficacy Study part: at least 7 moderate to severe bothersome VMS per day or at least 50 moderate to severe bothersome VMS per week in the last 7 consecutive days during the Screening period;
  2. For the Endometrial and General Safety Study part: at least 1 moderate to severe VMS per week;
* Body mass index ≥ 18.0 kg/m^2 to ≤ 38.0 kg/m^2;
* A mammogram that shows no sign of significant disease performed during screening or within 9 months prior to the start of screening ;
* Post-menopausal status defined as any of the following:
* For non-hysterectomized subjects:

  1. at least 12 months of spontaneous amenorrhea with serum follicle stimulating hormone (FSH) >40 milli-International unit (mIU)/mL (value obtained after washout of estrogen/progestin containing drugs, see exclusion criteria 18 and 20);
  2. or at least 6 months of spontaneous amenorrhea with serum FSH >40 mIU/mL and E2 <20 pg/mL (<73.4 pmol/L,value obtained after washout of estrogen/progestin containing drugs, see exclusion criteria 18 and 20);
  3. or at least 6 weeks postsurgical bilateral oophorectomy;
* For hysterectomized subjects:

  1. serum FSH >40 mIU/mL and E2 <20 pg/mL (<73.4 pmol/L, values obtained after washout of estrogen/progestin containing drug see exclusion criteria 18 and 20);
  2. or at least 6 weeks post-surgical bilateral oophorectomy.
* Good physical and mental health, in the judgement of the Investigator as based on medical history, physical and gynecological examination and clinical assessments performed prior Visit 1;
* Able to understand and comply with the protocol requirements, instructions, and protocol-stated restrictions;
* Able and willing to complete trial daily paper diaries (if applicable) and questionnaires.

Exclusion Criteria:

* History of malignancy with the exception of basal cell or squamous cell carcinoma of the skin if diagnosed more than 1 year prior to the Screening visit;
* Any clinically significant findings found by the Investigator at the breast examination and/or on mammography suspicious of breast malignancy that would require additional clinical testing to rule out breast cancer (however, simple cysts confirmed by ultrasound are allowed);
* Papanicolaou (PAP) test with atypical squamous cells undetermined significance (ASC-US) or higher (low-grade intraepithelial lesion [LSIL], atypical squamous cells- cannot exclude high-grade intraepithelial lesion [HSIL] [ASC-H], HSIL, dysplastic or malignant cells) in sub-totally hysterectomized and non-hysterectomized subjects . Note: ASC-US is allowed if a reflex human papilloma virus (HPV) testing is performed and is negative for high risk oncogene HPV subtypes 16 and 18;
* For non-hysterectomized subjects:

  1. History or presence of uterine cancer, endometrial hyperplasia, or disordered proliferative endometrium;
  2. Presence of endometrial polyps;
  3. Undiagnosed vaginal bleeding or undiagnosed abnormal uterine bleeding;
  4. Endometrial ablation;
  5. Any uterine/endometrial abnormality that in the judgment of the investigator contraindicates the use of estrogen and/or progestin therapy. This includes presence or history of adenomyosis or significant myoma;
* Systolic blood pressure (BP) higher than 130 mmHg, diastolic BP higher than 80 mmHg during screening;
* History of venous or arterial thromboembolic disease (e.g., superficial or deep vein thrombosis, pulmonary embolism, stroke, myocardial infarction, angina pectoris, etc.), or first degree family history of venous thromboembolism (VTE);
* History of known acquired or congenital coagulopathy or abnormal coagulation factors, including known thrombophilia's;
* Laboratory values of fasting glucose above 125 mg/dL (>6.94 mmol/L) and/or glycated hemoglobin above 7%18;
* Dyslipoproteinemia (LDL >190 mg/dL [>4.91 mmol/L] and/or triglycerides >300 mg/dL [>3.39 mmol/L])19;
* Subjects smoking >15 cigarettes per day;
* Presence or history of gallbladder disease, unless cholecystectomy has been performed;
* Systemic lupus erythematosus;
* Any malabsorption disorders including gastric by-pass surgery;
* History of acute liver disease in the preceding 12 months before the start of screening or presence or history of chronic or severe liver disease [alanine transaminase (ALT) or aspartate transaminase (AST) >2x upper limit of normal (ULN), bilirubin >1.5 ULN]; or liver tumors;
* Chronic or current acute renal impairment (estimated glomerular filtration rate <60 ml/min);
* Porphyria;
* Diagnosis or treatment of major psychiatric disorder (e.g., schizophrenia, bipolar disorder, etc.), in the judgement of the Investigator;
* Use of estrogen/progestin containing drug(s) up to:

  1. 1 week before screening start for vaginal non systemic hormonal products (rings, creams, gels);
  2. 4 weeks before screening start for vaginal or transdermal estrogen or estrogen/progestin products;
  3. 8 weeks before screening start for oral estrogen and/or progestin products and/or selective estrogen receptor modulator therapy;
  4. 8 weeks before screening start for intrauterine progestin therapy;
  5. 3 months before screening start for progestin implants or estrogen alone injectable drug therapy;
  6. 6 months before screening start for estrogen pellet therapy or progestin injectable drug therapy;
* Use of androgen/dehydroepiandrosterone (DHEA) containing drugs:

  1. 8 weeks before screening start for oral, topical, vaginal or transdermal androgen;
  2. 6 months before screening start for implantable or injectable androgen therapy;
* Use of phytoestrogens or black cohosh for the treatment of VMS up to 2 weeks before the start of screening;
* For the women participating in the Efficacy Study part: use of prescription or over-the-counter products used for the treatment of VMS, e.g., anti-depressants: paroxetine, escitalopram, methyldopa, opioid and clonidine up to 4 weeks before the start of screening, and venlafaxine and desvenlafaxine up to 3 months before the start of screening , and not willing to stop these during their participation in the trial;
* Not willing to stop any hormonal products as described in exclusion criteria 18, 19 and 20, during their participation in the trial;
* Inadequately treated hyperthyroidism with abnormal TSH and free T4 at screening. Subjects with low or high TSH are allowed if free T4 at screening is within normal range;
* History or presence of allergy/intolerance to the investigational product or drugs of this class or any component of it, or history of drug or other allergy that, in the opinion of the Investigator contraindicates subject participation;
* History of alcohol or substance abuse (including marijuana, even if legally allowed) or dependence in the previous 12 months before the start of screening as determined by the Investigator, based on reported observations;
* Sponsor or contract research organization (CRO) employees or employees under the direct supervision of the Investigator and/or involved directly in the trial;
* Subjects with known or suspected history of a clinically significant systemic disease, unstable medical disorders, life-threatening disease or current malignancies that would pose a risk to the subject in the opinion of the Investigator;
* Participation in another investigational drug clinical trial within 1 month (30 days) or having received an investigational drug within the last month (30 days) before the start of screening;
* Is judged by the Investigator to be unsuitable for any reason;
* For non-hysterectomized subjects to be included in the USA and Canada: history or presence of allergy to peanuts.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1570 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
Mean change in weekly frequency of moderate to severe vasomotor symptoms (VMS) from Baseline to Week 4 (Efficacy Study Part) | Baseline and Week 4
  The weekly frequency of moderate to severe VMS at Baseline and Week 4 is defined as the total number (sum) of all recorded moderate to severe VMS experienced during the last 7 consecutive days prior randomization for Baseline and at Week 4.
  Mean change = mean weekly frequency at Week 4 - mean weekly frequency at Baseline
Mean change in weekly frequency of moderate to severe vasomotor symptoms (VMS) from Baseline to Week 12 (Efficacy Study Part) | Baseline and Week 12
  The weekly frequency of moderate to severe VMS at Baseline and Week 12 is defined as the total number (sum) of all recorded moderate to severe VMS experienced during the last 7 consecutive days prior randomization for Baseline and at Week 12.
  Mean change = mean weekly frequency at Week 12 - mean weekly frequency at Baseline
Mean change in severity of moderate to severe vasomotor symptoms (VMS) from Baseline to Week 4 (Efficacy Study Part) | Baseline and Week 4
  The severity score is derived as follows: mild = 1, moderate = 2, and severe = 3.
  The mean severity score of VMS at Baseline and Week 4 is defined as the arithmetic mean of the daily severity score values of moderate and severe VMS observed from the last 7 days prior randomization for Baseline and of moderate and severe VMS observed at Week 4.
  Baseline and Week 4 severity score = [(2 x number of moderate VMS) + (3 x number of severe VMS)]/ (total number of moderate + severe VMS).
  Mean change = mean severity score at Week 4 - mean severity score at Baseline
Mean change in severity of moderate to severe vasomotor symptoms (VMS) from Baseline to Week 12 (Efficacy Study Part) | Baseline and Week 12
  The severity score is derived as follows: mild = 1, moderate = 2, and severe = 3.
  The mean severity score of VMS at Baseline and Week 12 is defined as the arithmetic mean of the daily severity score values of moderate and severe VMS observed from the last 7 days prior randomization for Baseline and of moderate and severe VMS observed at Week 12.
  Baseline and Week 12 severity score = [(2 x number of moderate VMS) + (3 x number of severe VMS)]/ (total number of moderate + severe VMS).
  Mean change = mean severity score at Week 12 - mean severity score at Baseline
Incidence of endometrial hyperplasia with up to 12 months of treatment based on endometrial biopsies (Endometrial and General Safety Study Part) | Screening and Week 53
  Endometrial biopsies will be centrally evaluated by three independent expert pathologists from different institutions, blinded to treatment group and to each other's readings. The concurrence of two of the three pathologists will be accepted as the final diagnosis. If there is no agreement among the three pathologists, the most severe pathologic diagnosis, i.e., atypical hyperplasia >complex hyperplasia >simple hyperplasia >benign endometrium, will be used as the final diagnosis.

SECONDARY OUTCOMES:
Mean change from Baseline to Week 1 in the weekly frequency and severity of moderate to severe vasomotor symptoms (VMS) (Efficacy Study Part) | Baseline and Week 1
  The weekly frequency of moderate to severe VMS at Baseline and Week 1 is defined as the total number (sum) of all recorded moderate to severe VMS experienced during the last 7 consecutive days prior randomization for Baseline and at Week 1.
  Mean change = mean weekly frequency at Week 1 - mean weekly frequency at Baseline
  The severity score is derived as follows: mild = 1, moderate = 2, and severe = 3.
  The mean severity score of VMS at Baseline and Week 1 is defined as the arithmetic mean of the daily severity score values of moderate and severe VMS observed from the last 7 days prior randomization for Baseline and of moderate and severe VMS observed at Week 1.
  Baseline and Week 1 severity score = [(2 x number of moderate VMS) + (3 x number of severe VMS)]/ (total number of moderate + severe VMS).
  Mean change = mean severity score at Week 1 - mean severity score at Baseline
Mean change from Baseline to Week 2 in the weekly frequency and severity of moderate to severe vasomotor symptoms (VMS) (Efficacy Study Part) | Baseline and Week 2
  The weekly frequency of moderate to severe VMS at Baseline and Week 2 is defined as the total number (sum) of all recorded moderate to severe VMS experienced during the last 7 consecutive days prior randomization for Baseline and at Week 2.
  Mean change = mean weekly frequency at Week 2 - mean weekly frequency at Baseline
  The severity score is derived as follows: mild = 1, moderate = 2, and severe = 3.
  The mean severity score of VMS at Baseline and Week 2 is defined as the arithmetic mean of the daily severity score values of moderate and severe VMS observed from the last 7 days prior randomization for Baseline and of moderate and severe VMS observed at Week 2.
  Baseline and Week 2 severity score = [(2 x number of moderate VMS) + (3 x number of severe VMS)]/ (total number of moderate + severe VMS).
  Mean change = mean severity score at Week 2 - mean severity score at Baseline
Mean change from Baseline to Week 3 in the weekly frequency and severity of moderate to severe vasomotor symptoms (VMS) ((Efficacy Study Part) | Baseline and Week 3
  The weekly frequency of moderate to severe VMS at Baseline and Week 3 is defined as the total number (sum) of all recorded moderate to severe VMS experienced during the last 7 consecutive days prior randomization for Baseline and at Week 3.
  Mean change = mean weekly frequency at Week 3 - mean weekly frequency at Baseline
  The severity score is derived as follows: mild = 1, moderate = 2, and severe = 3.
  The mean severity score of VMS at Baseline and Week 3 is defined as the arithmetic mean of the daily severity score values of moderate and severe VMS observed from the last 7 days prior randomization for Baseline and of moderate and severe VMS observed at Week 3.
  Baseline and Week 3 severity score = [(2 x number of moderate VMS) + (3 x number of severe VMS)]/ (total number of moderate + severe VMS).
  Mean change = mean severity score at Week 3 - mean severity score at Baseline
Mean change from Baseline to Week 4 in the weekly frequency and severity of moderate to severe vasomotor symptoms (VMS) (Efficacy part) | Baseline and Week 4
  The weekly frequency of moderate to severe VMS at Baseline and Week 4 is defined as the total number (sum) of all recorded moderate to severe VMS experienced during the last 7 consecutive days prior randomization for Baseline and at Week 4.
  Mean change = mean weekly frequency at Week 4 - mean weekly frequency at Baseline
  The severity score is derived as follows: mild = 1, moderate = 2, and severe = 3.
  The mean severity score of VMS at Baseline and Week 4 is defined as the arithmetic mean of the daily severity score values of moderate and severe VMS observed from the last 7 days prior randomization for Baseline and of moderate and severe VMS observed at Week 4.
  Baseline and Week 4 severity score = [(2 x number of moderate VMS) + (3 x number of severe VMS)]/ (total number of moderate + severe VMS).
  Mean change = mean severity score at Week 4 - mean severity score at Baseline
Mean change from Baseline to Week 5 in the weekly frequency and severity of moderate to severe vasomotor symptoms (VMS) (Efficacy Study Part) | Baseline and Week 5
  The weekly frequency of moderate to severe VMS at Baseline and Week 5 is defined as the total number (sum) of all recorded moderate to severe VMS experienced during the last 7 consecutive days prior randomization for Baseline and at Week 5.
  Mean change = mean weekly frequency at Week 5 - mean weekly frequency at Baseline
  The severity score is derived as follows: mild = 1, moderate = 2, and severe = 3.
  The mean severity score of VMS at Baseline and Week 5 is defined as the arithmetic mean of the daily severity score values of moderate and severe VMS observed from the last 7 days prior randomization for Baseline and of moderate and severe VMS observed at Week 5.
  Baseline and Week 5 severity score = [(2 x number of moderate VMS) + (3 x number of severe VMS)]/ (total number of moderate + severe VMS).
  Mean change = mean severity score at Week 5 - mean severity score at Baseline
Mean change from Baseline to Week 6 in the weekly frequency and severity of moderate to severe vasomotor symptoms (VMS) (Efficacy Study Part) | Baseline and Week 6
  The weekly frequency of moderate to severe VMS at Baseline and Week 6 is defined as the total number (sum) of all recorded moderate to severe VMS experienced during the last 7 consecutive days prior randomization for Baseline and at Week 6.
  Mean change = mean weekly frequency at Week 6 - mean weekly frequency at Baseline
  The severity score is derived as follows: mild = 1, moderate = 2, and severe = 3.
  The mean severity score of VMS at Baseline and Week 6 is defined as the arithmetic mean of the daily severity score values of moderate and severe VMS observed from the last 7 days prior randomization for Baseline and of moderate and severe VMS observed at Week 6.
  Baseline and Week 6 severity score = [(2 x number of moderate VMS) + (3 x number of severe VMS)]/ (total number of moderate + severe VMS).
  Mean change = mean severity score at Week 6 - mean severity score at Baseline
Mean change from Baseline to Week 7 in the weekly frequency and severity of moderate to severe vasomotor symptoms (VMS) (Efficacy Study Part) | Baseline and Week 7
  The weekly frequency of moderate to severe VMS at Baseline and Week 7 is defined as the total number (sum) of all recorded moderate to severe VMS experienced during the last 7 consecutive days prior randomization for Baseline and at Week 7.
  Mean change = mean weekly frequency at Week 7 - mean weekly frequency at Baseline
  The severity score is derived as follows: mild = 1, moderate = 2, and severe = 3.
  The mean severity score of VMS at Baseline and Week 7 is defined as the arithmetic mean of the daily severity score values of moderate and severe VMS observed from the last 7 days prior randomization for Baseline and of moderate and severe VMS observed at Week 7.
  Baseline and Week 7 severity score = [(2 x number of moderate VMS) + (3 x number of severe VMS)]/ (total number of moderate + severe VMS).
  Mean change = mean severity score at Week 7 - mean severity score at Baseline
Mean change from Baseline to Week 8 in the weekly frequency and severity of moderate to severe vasomotor symptoms (VMS) (Efficacy Study Part) | Baseline and Week 8
  The weekly frequency of moderate to severe VMS at Baseline and Week 8 is defined as the total number (sum) of all recorded moderate to severe VMS experienced during the last 7 consecutive days prior randomization for Baseline and at Week 8.
  Mean change = mean weekly frequency at Week 8 - mean weekly frequency at Baseline
  The severity score is derived as follows: mild = 1, moderate = 2, and severe = 3.
  The mean severity score of VMS at Baseline and Week 8 is defined as the arithmetic mean of the daily severity score values of moderate and severe VMS observed from the last 7 days prior randomization for Baseline and of moderate and severe VMS observed at Week 8.
  Baseline and Week 8 severity score = [(2 x number of moderate VMS) + (3 x number of severe VMS)]/ (total number of moderate + severe VMS).
  Mean change = mean severity score at Week 8 - mean severity score at Baseline
Mean change from Baseline to Week 9 in the weekly frequency and severity of moderate to severe vasomotor symptoms (VMS) (Efficacy Study Part) | Baseline and Week 9
  The weekly frequency of moderate to severe VMS at Baseline and Week 9 is defined as the total number (sum) of all recorded moderate to severe VMS experienced during the last 7 consecutive days prior randomization for Baseline and at Week 9.
  Mean change = mean weekly frequency at Week 9 - mean weekly frequency at Baseline
  The severity score is derived as follows: mild = 1, moderate = 2, and severe = 3.
  The mean severity score of VMS at Baseline and Week 9 is defined as the arithmetic mean of the daily severity score values of moderate and severe VMS observed from the last 7 days prior randomization for Baseline and of moderate and severe VMS observed at Week 9.
  Baseline and Week 9 severity score = [(2 x number of moderate VMS) + (3 x number of severe VMS)]/ (total number of moderate + severe VMS).
  Mean change = mean severity score at Week 9 - mean severity score at Baseline
Mean change from Baseline to Week 10 in the weekly frequency and severity of moderate to severe vasomotor symptoms (VMS) (Efficacy Study Part) | Baseline and Week 10
  The weekly frequency of moderate to severe VMS at Baseline and Week 10 is defined as the total number (sum) of all recorded moderate to severe VMS experienced during the last 7 consecutive days prior randomization for Baseline and at Week 10.
  Mean change = mean weekly frequency at Week 10 - mean weekly frequency at Baseline
  The severity score is derived as follows: mild = 1, moderate = 2, and severe = 3.
  The mean severity score of VMS at Baseline and Week 10 is defined as the arithmetic mean of the daily severity score values of moderate and severe VMS observed from the last 7 days prior randomization for Baseline and of moderate and severe VMS observed at Week 10.
  Baseline and Week 10 severity score = [(2 x number of moderate VMS) + (3 x number of severe VMS)]/ (total number of moderate + severe VMS).
  Mean change = mean severity score at Week 10 - mean severity score at Baseline
Mean change from Baseline to Week 11 in the weekly frequency and severity of moderate to severe vasomotor symptoms (VMS) (Efficacy Study Part) | Baseline and Week 11
  The weekly frequency of moderate to severe VMS at Baseline and Week 11 is defined as the total number (sum) of all recorded moderate to severe VMS experienced during the last 7 consecutive days prior randomization for Baseline and at Week 11.
  Mean change = mean weekly frequency at Week 11 - mean weekly frequency at Baseline
  The severity score is derived as follows: mild = 1, moderate = 2, and severe = 3.
  The mean severity score of VMS at Baseline and Week 11 is defined as the arithmetic mean of the daily severity score values of moderate and severe VMS observed from the last 7 days prior randomization for Baseline and of moderate and severe VMS observed at Week 11.
  Baseline and Week 11 severity score = [(2 x number of moderate VMS) + (3 x number of severe VMS)]/ (total number of moderate + severe VMS).
  Mean change = mean severity score at Week 11 - mean severity score at Baseline
Mean change from Baseline to Week 12 in the weekly frequency and severity of moderate to severe vasomotor symptoms (VMS) (Efficacy Study Part) | Baseline and Week 12
  The weekly frequency of moderate to severe VMS at Baseline and Week 12 is defined as the total number (sum) of all recorded moderate to severe VMS experienced during the last 7 consecutive days prior randomization for Baseline and at Week 12.
  Mean change = mean weekly frequency at Week 12 - mean weekly frequency at Baseline
  The severity score is derived as follows: mild = 1, moderate = 2, and severe = 3.
  The mean severity score of VMS at Baseline and Week 12 is defined as the arithmetic mean of the daily severity score values of moderate and severe VMS observed from the last 7 days prior randomization for Baseline and of moderate and severe VMS observed at Week 12.
  Baseline and Week 12 severity score = [(2 x number of moderate VMS) + (3 x number of severe VMS)]/ (total number of moderate + severe VMS).
  Mean change = mean severity score at Week 12 - mean severity score at Baseline
Mean change from Baseline to Week 1 in the weekly frequency and severity of mild, moderate and severe vasomotor symptoms (VMS) (Efficacy Study Part) | Baseline and Week 1
  The severity score is derived as follows: mild = 1, moderate = 2, and severe = 3.
  The mean severity score of VMS at Baseline and Week 1 is defined as the arithmetic mean of the daily severity score values of mild, moderate and severe VMS observed from the last 7 days prior randomization for Baseline and of mild, moderate and severe VMS observed at Week 1.
  Baseline and Week 1 severity score = [(1 x number of mild VMS) + (2 x number of moderate VMS) + (3 x number of severe VMS)]/ (total number of mild + moderate + severe VMS).
  Mean change = mean severity score at Week 1 - mean severity score at Baseline
Mean change from Baseline to Week 2 in the weekly frequency and severity of mild, moderate and severe vasomotor symptoms (VMS) (Efficacy Study Part) | Baseline and Week 2
  The severity score is derived as follows: mild = 1, moderate = 2, and severe = 3.
  The mean severity score of VMS at Baseline and Week 2 is defined as the arithmetic mean of the daily severity score values of mild, moderate and severe VMS observed from the last 7 days prior randomization for Baseline and of mild, moderate and severe VMS observed at Week 2.
  Baseline and Week 2 severity score = [(1 x number of mild VMS) + (2 x number of moderate VMS) + (3 x number of severe VMS)]/ (total number of mild + moderate + severe VMS).
  Mean change = mean severity score at Week 2 - mean severity score at Baseline
Mean change from Baseline to Week 3 in the weekly frequency and severity of mild, moderate and severe vasomotor symptoms (VMS) (Efficacy Study Part) | Baseline and Week 3
  The severity score is derived as follows: mild = 1, moderate = 2, and severe = 3.
  The mean severity score of VMS at Baseline and Week 3 is defined as the arithmetic mean of the daily severity score values of mild, moderate and severe VMS observed from the last 7 days prior randomization for Baseline and of mild, moderate and severe VMS observed at Week 3.
  Baseline and Week 3 severity score = [(1 x number of mild VMS) + (2 x number of moderate VMS) + (3 x number of severe VMS)]/ (total number of mild + moderate + severe VMS).
  Mean change = mean severity score at Week 3 - mean severity score at Baseline
Mean change from Baseline to Week 4 in the weekly frequency and severity of mild, moderate and severe vasomotor symptoms (VMS) (Efficacy Study Part) | Baseline and Week 4
  The severity score is derived as follows: mild = 1, moderate = 2, and severe = 3.
  The mean severity score of VMS at Baseline and Week 4 is defined as the arithmetic mean of the daily severity score values of mild, moderate and severe VMS observed from the last 7 days prior randomization for Baseline and of mild, moderate and severe VMS observed at Week 4.
  Baseline and Week 4 severity score = [(1 x number of mild VMS) + (2 x number of moderate VMS) + (3 x number of severe VMS)]/ (total number of mild + moderate + severe VMS).
  Mean change = mean severity score at Week 4 - mean severity score at Baseline
Mean change from Baseline to Week 5 in the weekly frequency and severity of mild, moderate and severe vasomotor symptoms (VMS) (Efficacy Study Part) | Baseline and Week 5
  The severity score is derived as follows: mild = 1, moderate = 2, and severe = 3.
  The mean severity score of VMS at Baseline and Week 5 is defined as the arithmetic mean of the daily severity score values of mild, moderate and severe VMS observed from the last 7 days prior randomization for Baseline and of mild, moderate and severe VMS observed at Week 5.
  Baseline and Week 5 severity score = [(1 x number of mild VMS) + (2 x number of moderate VMS) + (3 x number of severe VMS)]/ (total number of mild + moderate + severe VMS).
  Mean change = mean severity score at Week 5 - mean severity score at Baseline
Mean change from Baseline to Week 6 in the weekly frequency and severity of mild, moderate and severe vasomotor symptoms (VMS) (Efficacy Study Part) | Baseline and Week 6
  The severity score is derived as follows: mild = 1, moderate = 2, and severe = 3.
  The mean severity score of VMS at Baseline and Week 6 is defined as the arithmetic mean of the daily severity score values of mild, moderate and severe VMS observed from the last 7 days prior randomization for Baseline and of mild, moderate and severe VMS observed at Week 6.
  Baseline and Week 6 severity score = [(1 x number of mild VMS) + (2 x number of moderate VMS) + (3 x number of severe VMS)]/ (total number of mild + moderate + severe VMS).
  Mean change = mean severity score at Week 6 - mean severity score at Baseline
Mean change from Baseline to Week 7 in the weekly frequency and severity of mild, moderate and severe vasomotor symptoms (VMS) (Efficacy Study Part) | Baseline and Week 7
  The severity score is derived as follows: mild = 1, moderate = 2, and severe = 3.
  The mean severity score of VMS at Baseline and Week 7 is defined as the arithmetic mean of the daily severity score values of mild, moderate and severe VMS observed from the last 7 days prior randomization for Baseline and of mild, moderate and severe VMS observed at Week 7.
  Baseline and Week 7 severity score = [(1 x number of mild VMS) + (2 x number of moderate VMS) + (3 x number of severe VMS)]/ (total number of mild + moderate + severe VMS).
  Mean change = mean severity score at Week 7 - mean severity score at Baseline
Mean change from Baseline to Week 8 in the weekly frequency and severity of mild, moderate and severe vasomotor symptoms (VMS) (Efficacy Study Part) | Baseline and Week 8
  The severity score is derived as follows: mild = 1, moderate = 2, and severe = 3.
  The mean severity score of VMS at Baseline and Week 8 is defined as the arithmetic mean of the daily severity score values of mild, moderate and severe VMS observed from the last 7 days prior randomization for Baseline and of mild, moderate and severe VMS observed at Week 8.
  Baseline and Week 8 severity score = [(1 x number of mild VMS) + (2 x number of moderate VMS) + (3 x number of severe VMS)]/ (total number of mild + moderate + severe VMS).
  Mean change = mean severity score at Week 8 - mean severity score at Baseline
Mean change from Baseline to Week 9 in the weekly frequency and severity of mild, moderate and severe vasomotor symptoms (VMS) (Efficacy Study Part) | Baseline and Week 9
  The severity score is derived as follows: mild = 1, moderate = 2, and severe = 3.
  The mean severity score of VMS at Baseline and Week 9 is defined as the arithmetic mean of the daily severity score values of mild, moderate and severe VMS observed from the last 7 days prior randomization for Baseline and of mild, moderate and severe VMS observed at Week 9.
  Baseline and Week 9 severity score = [(1 x number of mild VMS) + (2 x number of moderate VMS) + (3 x number of severe VMS)]/ (total number of mild + moderate + severe VMS).
  Mean change = mean severity score at Week 9 - mean severity score at Baseline
Mean change from Baseline to Week 10 in the weekly frequency and severity of mild, moderate and severe vasomotor symptoms (VMS) (Efficacy Study Part) | Baseline and Week 10
  The severity score is derived as follows: mild = 1, moderate = 2, and severe = 3.
  The mean severity score of VMS at Baseline and Week 10 is defined as the arithmetic mean of the daily severity score values of mild, moderate and severe VMS observed from the last 7 days prior randomization for Baseline and of mild, moderate and severe VMS observed at Week 10.
  Baseline and Week 10 severity score = [(1 x number of mild VMS) + (2 x number of moderate VMS) + (3 x number of severe VMS)]/ (total number of mild + moderate + severe VMS).
  Mean change = mean severity score at Week 10 - mean severity score at Baseline
Mean change from Baseline to Week 11 in the weekly frequency and severity of mild, moderate and severe vasomotor symptoms (VMS) (Efficacy Study Part) | Baseline and Week 11
  The severity score is derived as follows: mild = 1, moderate = 2, and severe = 3.
  The mean severity score of VMS at Baseline and Week 11 is defined as the arithmetic mean of the daily severity score values of mild, moderate and severe VMS observed from the last 7 days prior randomization for Baseline and of mild, moderate and severe VMS observed at Week 11.
  Baseline and Week 11 severity score = [(1 x number of mild VMS) + (2 x number of moderate VMS) + (3 x number of severe VMS)]/ (total number of mild + moderate + severe VMS).
  Mean change = mean severity score at Week 11 - mean severity score at Baseline
Mean change from Baseline to Week 12 in the weekly frequency and severity of mild, moderate and severe vasomotor symptoms (VMS) (Efficacy Study Part) | Baseline and Week 12
  The severity score is derived as follows: mild = 1, moderate = 2, and severe = 3.
  The mean severity score of VMS at Baseline and Week 12 is defined as the arithmetic mean of the daily severity score values of mild, moderate and severe VMS observed from the last 7 days prior randomization for Baseline and of mild, moderate and severe VMS observed at Week 12.
  Baseline and Week 12 severity score = [(1 x number of mild VMS) + (2 x number of moderate VMS) + (3 x number of severe VMS)]/ (total number of mild + moderate + severe VMS).
  Mean change = mean severity score at Week 12 - mean severity score at Baseline
Percentage of participants with 50% reduction from Baseline in the weekly frequency of moderate to severe vasomotor symptoms (VMS) at Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 (Efficacy Study Part) | Baseline, Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12
  The weekly frequency of moderate to severe VMS at Baseline and Week X is defined as the total number (sum) of all recorded moderate to severe VMS experienced during the last 7 consecutive days prior randomization (Baseline) and day [(X-1)*7+1] to day X*7 (Week X).
Percentage of participants with 50% reduction from Baseline in the weekly frequency of mild, moderate, and severe vasomotor symptoms (VMS) at Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 (Efficacy Study Part) | Baseline, Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12
  The weekly frequency of moderate to severe VMS at Baseline and Week X is defined as the total number (sum) of all recorded moderate to severe VMS experienced during the last 7 consecutive days prior randomization (Baseline) and day [(X-1)*7+1] to day X*7 (Week X).
Percentage of participants with 75% reduction from Baseline in the weekly frequency of moderate to severe VMS at Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 (Efficacy Study Part) | Baseline, Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12
  The weekly frequency of moderate to severe VMS at Baseline and Week X is defined as the total number (sum) of all recorded moderate to severe VMS experienced during the last 7 consecutive days prior randomization (Baseline) and day [(X-1)*7+1] to day X*7 (Week X).
Percentage of participants with 75% reduction from Baseline in the weekly frequency of mild, moderate, and severe VMS at Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 (Efficacy Study Part) | Baseline, Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12
  The weekly frequency of moderate to severe VMS at Baseline and Week X is defined as the total number (sum) of all recorded moderate to severe VMS experienced during the last 7 consecutive days prior randomization (Baseline) and day [(X-1)*7+1] to day X*7 (Week X).
Percentage of participants with a clinically important difference (CID) compared to Baseline in the weekly frequency of moderate to severe VMS at Week 4 using the Clinical Global Impression (CGI) questionnaire (Efficacy Study Part) | Week 4
  The CGI score is a seven point scale in which subjects will be asked to rate the total improvement, whether or not in her judgment it was due entirely to drug treatment, compared to her condition at admission to the study. Scale: Very much improved, Much improved, Minimally improved, No change, Minimally worse, Much worse, Very much worse.
Percentage of participants with a clinically important difference (CID) compared to baseline in the weekly frequency of moderate to severe VMS at Week 12 using the Clinical Global Impression (CGI) questionnaire (Efficacy Study Part) | Week 12
  The CGI score is a seven point scale in which subjects will be asked to rate the total improvement, whether or not in her judgment it was due entirely to drug treatment, compared to her condition at admission to the study. Scale: Very much improved, Much improved, Minimally improved, No change, Minimally worse, Much worse, Very much worse.
Change from Baseline to Week 12 in vulvovaginal atrophy (VVA) symptoms (Efficacy Study Part) | Baseline and Week 12
  Genitourinary syndrome of menopause (GSM) will be assessed by the subjects using the vulvovaginal atrophy (VVA) self assessment questionnaire. The following GSM symptoms will be assessed:
  * Vaginal dryness
  * Vaginal and/or vulvar irritation/itching
  * Dysuria
  * Vaginal pain associated with sexual activity
  * Vaginal bleeding associated with sexual activity
  All GSM symptoms except vaginal bleeding associated with sexual activity will be graded by the participants using the following scale: [0] none, [1] mild, [2] moderate, or [3] severe. Vaginal bleeding associated with sexual activity is documented using 2 categories: [0] absent or [1] present. A negative change from baseline score indicates improvement in symptoms.
Change from Baseline to Week 12 in the vulvovaginal atrophy (VVA) symptom that is initially identified by the participant as being the most bothersome using the VVA questionnaire at baseline (Efficacy Study Part) | Baseline and Week 12
  Genitourinary syndrome of menopause (GSM) will be assessed by the subjects using the vulvovaginal atrophy (VVA) self assessment questionnaire. The following GSM symptoms will be assessed:
  * Vaginal dryness
  * Vaginal and/or vulvar irritation/itching
  * Dysuria
  * Vaginal pain associated with sexual activity
  * Vaginal bleeding associated with sexual activity
  All GSM symptoms except vaginal bleeding associated with sexual activity were graded by the participants using the following scale: [0] none, [1] mild, [2] moderate, or [3] severe. Vaginal bleeding associated with sexual activity was documented using 2 categories: [0] absent or [1] present. A negative change from baseline score indicates improvement in symptoms.
  At baseline the participant will be asked which of the above mentioned symptoms she identifies as being the most bothersome.
Change from Baseline to Week 12 in plasma concentration of triglycerides (Efficacy Study Part) | Baseline and Week 12
Change from Baseline to Week 12 in plasma concentration of low-density lipoprotein (LDL)-cholesterol (Efficacy Study Part) | Baseline and Week 12
Change from Baseline to Week 12 in plasma concentration of total cholesterol (Efficacy Study Part) | Baseline and Week 12
Change from Baseline to Week 12 in the total cholesterol/high density cholesterol (HDL) cholesterol ratio (Efficacy Study Part) | Baseline and Week 12
Change from Baseline to Week 12 in the HDL-cholesterol ratio (Efficacy Study Part) | Baseline and Week 12
Change from Baseline to Week 12 in plasma concentration of lipoprotein (a) (Efficacy Study Part) | Baseline and Week 12
Change from Baseline to Week 12 in fasting glycaemia (Efficacy Study part) | Baseline and Week 12
Change from Baseline to Week 12 in plasma concentration of insulin (Efficacy Study Part) | Baseline and Week 12
Change from Baseline to Week 12 in plasma concentration of glycated hemoglobin (Efficacy Study Part) | Baseline and Week 12
Change from Baseline to Week 12 in Homeostasis model-assessment-estimated insulin resistance (HOMA-IR) (Efficacy Study Part) | Baseline and Week 12
Change from baseline to Week 12 in health-related quality of life assessment (HRQoL) using the menopause-specific Quality of Life (MENQOL) questionnaire (Efficacy Study Part) | Baseline and Week 12
  The MENQOL is self-administered questionnaire which will assess changes in quality of life over a one-month period. It is composed of 29 questions indicating if subject experienced the problem (Yes/No) and if Yes, rating scale ranged from 0=Not bothered at all to 6=Extremely bothered. For analysis, the original scores will be converted to the analysis score ranging from 1-8 where No=1, 0=2, 1=3...and 6=8. The scale contains four domains: vasomotor, psychosocial, physical and sexual. Each domain is scored separately. Vasomotor domain score is mean of = Q1,Q2, Q3, with 1 being "not at all bothered" and 8 being "extremely bothered".
Total score in treatment satisfaction using the Clinical Global Impression (CGI) questionnaire (Efficacy Study Part) | Weeks 4 and 12
  The CGI score is a seven point scale in which subjects will be asked to rate the total improvement, whether or not in her judgment it was due entirely to drug treatment, compared to her condition at admission to the study. Scale: Very much improved, Much improved, Minimally improved, No change, Minimally worse, Much worse, Very much worse.
Number of participants with treatment-emergent adverse events (TEAEs) (Efficacy Study Part) | From baseline to Follow-up visit (up to Week 16)
  TEAEs are those adverse events occurring from time point of first ingestion of investigational product until last visit or any event already present that worsens in either intensity or frequency following exposure to the treatment.
Number of participants with changes in physical and gynecological examination results (Efficacy Study Part) | Screening and Week 13
  Physical examination will include an examination of general appearance, head, eyes, ears, nose, throat, skin, neck, lungs, breast, lymph nodes, abdomen, and the cardiovascular musculoskeletal and neurological systems.
  Gynecological examination will include a manual pelvic examination.
Number of participants with changes in vital sign results (Efficacy Study Part) | From screening to Week 13
  Vital signs will include height, body weight, body mass index, sitting systolic and diastolic blood pressures, and heart rate.
Number of participants with changes in electrocardiogram (ECG) results (Efficacy Study Part) | Screening and Week 13
  The ECG interpretation scheme will include the analysis of the morphology, rhythm, conduction, ST segment, PR, QRS, QT and corrected QT (QTc) intervals, T waves, U waves and the presence or absence of any pathological changes.
Number of participants with changes in breast examination results (Efficacy Study Part) | Screening and Week 13
Number of participants with changes in routine clinical laboratory test results (Efficacy Study Part) | Screening, Baseline and Week 13
  Routine laboratory tests include hematology and chemistry.
Change from baseline to each measured time point in endometrial thickness (Efficacy Study Part) | Screening, Week 13, Week 16
  Endometrial thickness will be assessed by transvaginal ultrasound (TVUS).
  Baseline: data will be recorded at Screening.
Frequency of subjects in the different endometrial categories according to Blaustein's pathology (Efficacy Study Part) | Screening and Week 13
  Endometrial biopsies will be centrally evaluated by three independent expert pathologists from different institutions, blinded to treatment group and to each other's readings. The concurrence of two of the three pathologists will be accepted as the final diagnosis. If there is no agreement among the three pathologists, the most severe pathologic diagnosis, i.e., atypical hyperplasia >complex hyperplasia >simple hyperplasia >benign endometrium, will be used as the final diagnosis.
Number of participants with vaginal bleeding and/or spotting during each 28-day cycle of treatment with E4 (Efficacy Study Part) | From Baseline up to Follow-up (Week 16)
  Vaginal bleeding will be daily recorded by the participant on the diary. Absence or occurrence of vaginal bleeding/ spotting will be assessed using the scale below: 0 = Absence of vaginal bleeding or spotting; 1 = Spotting: evidence of minimal blood loss requiring none or at most one pad, tampon or panty liner per day; 2 = Bleeding: evidence of blood loss requiring more than one pad, tampon or panty liner per day.
Number of days with bleeding and/or spotting during each 28-day cycle of treatment (Efficacy Study Part) | From Baseline up to Follow-up (Week 16)
  Vaginal bleeding will be daily recorded by the participant on the diary. Absence or occurrence of vaginal bleeding/spotting will be assessed using the scale below: 0 = Absence of vaginal bleeding or spotting; 1 = Spotting: evidence of minimal blood loss requiring none or at most one pad, tampon or panty liner per day; 2 = Bleeding: evidence of blood loss requiring more than one pad, tampon or panty liner per day.
Number of participants with amenorrhea (absence of any bleeding or spotting) during each 28-day cycle of treatment with E4 (Efficacy Study Part) | From Baseline up to Follow-up (Week 16)
  Vaginal bleeding will be daily recorded by the participant on the diary. Absence or occurrence of vaginal bleeding/ spotting will be assessed using the scale below: 0 = Absence of vaginal bleeding or spotting; 1 = Spotting: evidence of minimal blood loss requiring none or at most one pad, tampon or panty liner per day; 2 = Bleeding: evidence of blood loss requiring more than one pad, tampon or panty liner per day.
Cumulative rates of amenorrhea (Efficacy Study Part) | From Baseline up to Follow-up (Week 16)
  The rate of amenorrhea is defined as the percentage of women who reported consecutive cycles of amenorrhea for a given cycle of time.
Number of participants with treatment-emergent adverse events (TEAEs) (Endometrial and General Safety Part) | From baseline to Week 53
  TEAEs are those adverse events occurring from time point of first ingestion of investigational product until last visit or any event already present that worsens in either intensity or frequency following exposure to the treatment.
Number of participants with changes in physical and gynecological examination results (Endometrial and General Safety Part) | Screening and Week 53
  Physical examination will include an examination of general appearance, head, eyes, ears, nose, throat, skin, neck, lungs, breast, lymph nodes, abdomen, and the cardiovascular musculoskeletal and neurological systems.
  Gynecological examination will include a manual pelvic examination.
Number of participants with changes in vital sign results (Endometrial and General Safety Part) | From screening to Week 53
  Vital signs will include height, body weight, body mass index, sitting systolic and diastolic blood pressures, and heart rate.
Number of participants with changes in breast examination results (Endometrial and General Safety Part) | From screening to Week 53
  Vital signs will include height, body weight, body mass index, sitting systolic and diastolic blood pressures, and heart rate.
Number of participants with changes in electrocardiogram (ECG) results (Endometrial and General Safety Part) | Screening and Week 53
  The ECG interpretation scheme will include the analysis of the morphology, rhythm, conduction, ST segment, PR, QRS, QT and corrected QT (QTc) intervals, T waves, U waves and the presence or absence of any pathological changes.
Number of participants with changes in mammography results (Endometrial and General Safety Part) | Screening and Week 53
Number of participants with changes in routine clinical laboratory test results (Endometrial and General Safety Part) | Screening, Baseline and Week 13
  Routine laboratory tests include hematology and chemistry.
Number of women with vaginal bleeding and/or spotting during each 28-day cycle of treatment with E4 (Endometrial and General Safety Part) | From Baseline to Week 53
  Vaginal bleeding will be daily recorded by the participant on the diary. Absence or occurrence of vaginal bleeding/spotting will be assessed using the scale below: 0 = Absence of vaginal bleeding or spotting; 1 = Spotting: evidence of minimal blood loss requiring none or at most one pad, tampon or panty liner per day; 2 = Bleeding: evidence of blood loss requiring more than one pad, tampon or panty liner per day.
Number of days with bleeding and/or spotting during each 28-day cycle of treatment (Endometrial and General Safety Part) | From Baseline to Week 53
  Vaginal bleeding will be daily recorded by the participant on the diary. Absence or occurrence of vaginal bleeding/spotting will be assessed using the scale below: 0 = Absence of vaginal bleeding or spotting; 1 = Spotting: evidence of minimal blood loss requiring none or at most one pad, tampon or panty liner per day; 2 = Bleeding: evidence of blood loss requiring more than one pad, tampon or panty liner per day.
Number of participants with amenorrhea (absence of any bleeding or spotting) during each 28-day cycle of treatment with E4 (Endometrial and General Safety Part) | From Baseline to Week 53
  Vaginal bleeding will be daily recorded by the participant on the diary. Absence or occurrence of vaginal bleeding/spotting will be assessed using the scale below: 0 = Absence of vaginal bleeding or spotting; 1 = Spotting: evidence of minimal blood loss requiring none or at most one pad, tampon or panty liner per day; 2 = Bleeding: evidence of blood loss requiring more than one pad, tampon or panty liner per day.
Cumulative rates of amenorrhea (Endometrial and General Safety Part) | From Baseline to Week 53
  The rate of amenorrhea is defined as the percentage of women who reported consecutive cycles of amenorrhea for a given cycle of time.
Change from Baseline to Weeks 12 and 52 in health-related quality of life assessment (HRQoL) using the menopause-specific Quality of Life (MENQOL) questionnaire (Endometrial and General Safety Part) | Baseline and Weeks 12 and 52
  The MENQOL is self-administered questionnaire which will assess changes in quality of life over a one-month period. It is composed of 29 questions indicating if subject experienced the problem (Yes/No) and if Yes, rating scale ranged from 0=Not bothered at all to 6=Extremely bothered. For analysis, the original scores were converted to the analysis score ranging from 1-8 where No=1, 0=2, 1=3...and 6=8. The scale contains four domains: vasomotor, psychosocial, physical and sexual. Each domain is scored separately. Vasomotor domain score is mean of = Q1,Q2, Q3, with 1 being "not at all bothered" and 8 being "extremely bothered".
Total score in treatment satisfaction assessed after 4, 12 and 52 weeks of treatment using the Clinical Global Impression (CGI) questionnaire (Endometrial and General Safety Part) | Weeks 4, 12, and 52
  The CGI score is a seven point scale in which subjects will be asked to rate the total improvement, whether or not in her judgment it was due entirely to drug treatment, compared to her condition at admission to the study. Scale: Very much improved, Much improved, Minimally improved, No change, Minimally worse, Much worse, Very much worse.
Change from Baseline to Weeks 12 and 52 in plasma concentration of triglycerides (Endometrial and General Safety Part) | Baseline and Weeks 12 and 52
Change from Baseline to Weeks 12 and 52 in plasma concentration of high-density lipoprotein (HDL)-cholesterol (Endometrial and General Safety Part) | Baseline and Weeks 12 and 52
Change from Baseline to Weeks 12 and 52 in plasma concentration of low-density lipoprotein (LDL)-cholesterol (Endometrial and General Safety Part) | Baseline and Weeks 12 and 52
Change from Baseline to Weeks 12 and 52 in plasma concentration of total cholesterol (Endometrial and General Safety Part) | Baseline and Weeks 12 and 52
Change from Baseline to Weeks 12 and 52 in the total cholesterol/high density cholesterol (HDL) cholesterol ratio (Endometrial and General Safety Part) | Baseline and Weeks 12 and 52
Change from Baseline to Weeks 12 and 52 in plasma concentration of lipoprotein (a) (Endometrial and General Safety Part) | Baseline and Weeks 12 and 52
Change from Baseline to Weeks 12 and 52 in fasting glycaemia (Endometrial and General Safety Part) | Baseline and Weeks 12 and 52
Change from Baseline to Weeks 12 and 52 in plasma concentration of insulin (Endometrial and General Safety Part) | Baseline and Weeks 12 and 52
Change from Baseline to Weeks 12 and 52 in plasma concentration of glycated hemoglobin (Endometrial and General Safety Part) | Baseline and Weeks 12 and 52
Change from Baseline to Weeks 12 and 52 in Homeostasis model-assessment-estimated insulin resistance (HOMA-IR) (Endometrial and General Safety Part) | Baseline and Weeks 12 and 52
Change from Baseline to each measured time point in endometrial thickness (Endometrial and General Safety Study Part) | Screening, Baseline, Weeks 13, 29, and 53
  Endometrial thickness will be assessed by transvaginal ultrasound (TVUS).
Frequency of subjects in the different endometrial categories according to Blaustein's pathology (Endometrial and General Safety Study Part) | Screening and Week 53
  Endometrial biopsies will be centrally evaluated by three independent expert pathologists from different institutions, blinded to treatment group and to each other's readings. The concurrence of two of the three pathologists will be accepted as the final diagnosis. If there is no agreement among the three pathologists, the most severe pathologic diagnosis, i.e., atypical hyperplasia >complex hyperplasia >simple hyperplasia >benign endometrium, will be used as the final diagnosis.

CONTACTS AND LOCATIONS:
Locations (219):
- United States (62):
  - Estetra Study Site, Birmingham, Alabama
  - Estetra Study Site, Mesa, Arizona
  - Estetra Study Site, Phoenix, Arizona
  - Precision Trials AZ, LLC, Phoenix, Arizona
  - Noble Clinical Research, Tucson, Arizona
  - Hope Clinical Research, LLC, Canoga Park, California
  - Estetra Study Site, Pomona, California
  - Clinical Trials Research, Sacramento, California
  - Estetra Study Site, Sacramento, California
  - Estetra Study Site, Thousand Oaks, California
  - Estetra Study Site, West Covina, California
  - Velocity Clinical Research, Denver, Colorado
  - Estetra Study Site, Altamonte Springs, Florida
  - Estetra Study Site, Coconut Creek, Florida
  - Estetra Study Site, Hialeah, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Altus Research, Lake Worth, Florida
  - Medical Research Center of Miami II, Miami, Florida
  - Miami Clinical Research, Miami, Florida
  - Genoma Research Group, Inc., Miami, Florida
  - Estetra Study Site, Miami, Florida
  - San Marcus Research Clinic, Inc., Miami Lakes, Florida
  - Estetra Study Site, New Port Richey, Florida
  - Estetra Study Site, North Miami, Florida
  - Estetra Study Site, Ocoee, Florida
  - Clinical Neurosciecne Solutions, Inc. dba CNS Healthcare, Orlando, Florida
  - Estetra Study Site, Ormond Beach, Florida
  - Estetra Study Site, Palm Harbor, Florida
  - Estetra Study Site, Pembroke Pines, Florida
  - Estetra Study Site, Pinellas Park, Florida
  - Estetra Study Site, Port Saint Lucie, Florida
  - Physician Care Clinical Research, LLC, Sarasota, Florida
  - Estetra Study Site, Tampa, Florida
  - Estetra Study Site, Atlanta, Georgia
  - Infinite Clinical Trials, Morrow, Georgia
  - Fellows Research Alliance, Inc., Savannah, Georgia
  - Clinical Research Prime, Idaho Falls, Idaho
  - Praetorian Pharmaceutical Research, Marrero, Louisiana
  - Meridian Clinical Research, Norfolk, Nebraska
  - Jubilee Clinical Research, Inc, Las Vegas, Nevada
  - Excel Clinical Research, Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Bosque Women's Care, Albuquerque, New Mexico
  - PMG Research of Charlotte, LLC, Charlotte, North Carolina
  - Estetra Study Site, Durham, North Carolina
  - Estetra Study Site, Columbus, Ohio
  - Estetra Study Site, Englewood, Ohio
  - Estetra Study Site, Philadelphia, Pennsylvania
  - Magnolia Ob/Gyn Research Center, Myrtle Beach, South Carolina
  - Estetra Study Site, Chattanooga, Tennessee
  - Cedar Health Research, LLC, Dallas, Texas
  - Signature Gyn Services, Fort Worth, Texas
  - Estetra Study Site, Houston, Texas
  - Biopharma Informatic, Inc. Research Center, Houston, Texas
  - Cedar Health Research LLC, Irving, Texas
  - Estetra Study Site, Plano, Texas
  - Estetra Study Site, San Antonio, Texas
  - Estetra Study Site, Pleasant Grove, Utah
  - Estetra Study Site, Norfolk, Virginia
  - Tidewater Clinical Research Inc, Virginia Beach, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - IMA Clinical Research, Morgantown, West Virginia
- Argentina (9):
  - IDIM - Instituto de Investigaciones Metabolicas, Buenos Aires
  - Mautalen Salud e Investigacion, Buenos Aires
  - Fundacion Respirar (Centro Medico Dra. De Salvo) - Instituto Argentino de Investigaciones Clinicas (IAIC) S.R.L, Buenos Aires
  - Glenny Corp. S. A. / Bioclinica Argentina, Buenos Aires
  - Centro Medico Dra Laura Maffei Investigacion Clinica Aplicada, Caba
  - Centro de Investigacion Medico Lanus-CIMEL, Lanús
  - Centro De Investigaciones Medicas Mar Del Plata, Mar del Plata
  - Instituto de Investigaciones Clinicas Mar del Plata, Mar del Plata
  - Instituto Medico de la Fundacion Estudios Clinicos, Rosario
- Brazil (25):
  - Centro De Medicina Reprodutiva Ltda - Clinica Origen, Belo Horizonte
  - Faculdade de Medicina de Botucatu - UNESP, Botucatu
  - Centro De Pesquisa Clinica Do Brasil, Brasília
  - IPCC-Instituto de Pesquisa Clinica de Campinas, Campinas
  - University of Campinas Medical School, Campinas
  - Centro de Oncologia de Santa Catarina Ltda / Supera Oncologia, Chapecó
  - Instituto Tropical de Medicina Reprodutiva - Clinica INTRO, Cuiabá
  - CEPEME / CERHFAC Centro De Estudos E Pesquisas Em Reproducao Humana E Fertilizacao Assistida De Curitiba Ltda, Curitiba
  - Federal University Of Ceara, Fortaleza
  - Universidade Federal Do Rio Grande Do Norte/ Maternidade Escola Januario Cicco, Natal
  - Hospital Sao Vicente de Paulo, Associacao Hospitalar Beneficente Sao Vicente de Paulo, Passo Fundo
  - Hospital de Clinicas de Porto Alegre (HCPA), Porto Alegre
  - Nucleo de Pesquisa Clinica do Rio Grande do Sul Ltda, Porto Alegre
  - Unidade de Pesquisa Clínica - Centro de Medicina Reprodutiva, Porto Alegre
  - Hospital Sao Lucas da PUC, Porto Alegre
  - lnstituto Brasil De Pesquisa Clinica S.A (IBPCLIN), Rio de Janeiro
  - CEMEC - Faculdade de Medicina do ABC, São Bernardo do Campo
  - CPQuali Pesquisa Clinica LTDA, São Paulo
  - CPClin- Centro de Pesquisas Clinicas Ltda./Clinica Dr. Freddy Goldberg Eliaschewitz, São Paulo
  - Hospital Perola Byington/ Centro de Referencia da Saude da Mulher, São Paulo
  - Universidade Federal De Sao Paulo (Unifesp) - Hospital Sao Paulo (Hsp), São Paulo
  - CEPIC - Centro Paulista de Investigacao Clinica e Servicos Medicos Ltda, São Paulo
  - College - Centro De Pesquisa Clinica E Servicos Medicos Ltda College - Centro De Pesquisa Clinica (Baby Center Medicina Reprodutiva), São Paulo
  - CEDOES - Centro de Diagnostico e Pesquisa da Osteoporose do Espirito Santo, Vitória
  - Santa Casa De Votuporanga-Philanthropic hospital, Votuporanga
- Canada (9):
  - Aggarwal and Associates Limited, Brampton
  - DIEX Research Quebec, Québec
  - Clinique Rsf Inc., Québec
  - Estetra Study Site, Québec
  - Alpha Recherche Clinique, Québec
  - Estetra Study Site, Sarnia
  - Diex Research Sherbrooke Inc., Sherbrooke
  - Diex Recherche, Victoriaville
  - Fadia El Boreky Medicine Professional Corporation, Waterloo
- Czechia (21):
  - Dr. Vladimir Dvorak MD, Office Of, Brno
  - Gynekologie Meda Brno, Brno
  - Gynekologie Cheb s.r.o., Cheb
  - MUDr. Petr Sak, České Budějovice
  - Dr. Jiri Tiser MD, Office of, České Budějovice
  - GYN-Mika s.r.o., České Budějovice
  - MUDr. Martin Stepan s.r.o., Hradec Králové
  - Gynekologie Jihlava, Jihlava
  - MUDr. Jan Kestranek - gynekologicka ambulance, Náchod
  - Estetra Study Site, Olomouc
  - G-CENTRUM Olomouc, s.r.o., Olomouc
  - NEUMED gynekologicka ambulance s.r.o., Olomouc
  - Dr. Karel Buchta MD, Office of, Ostrava
  - Dr. Martina Maresova Rosenbergova MD, Office of, Pilsen
  - Gynekologicka ambulance Gyncare MUDr. Michael Svec s.r.o., Pilsen
  - Mediva s.r.o, Prague
  - Gynekologicko-porodnicka klinika, Prague
  - Dr. Lubomir Mikulasek, MD office Of, Prague
  - Vestra Clinics, Rychnov nad Kněžnou
  - Dr. Tereza Smrhova-Kovacs MD, Office of, Tábor
  - Dr. Ivana Salamonova MD, Office of, Vysoké
- Hungary (4):
  - Szent Anna Privat Surgery-Szent Anna Maganrendelo, Debrecen
  - Pecsi Tudomanyegyetem (PTE) Altalanos Orvostudomanyi Kar (AOK) - Klinikai Kozpont Szuleszeti es Nogyogyaszati Klinika, Pécs
  - Univ. of Szeged Faculty of General Medicine Albert Szent-Gyaergyi, Szeged
  - Csongrad Megyei Dr. Bugyi Istvan Korhaz, Szentes
- Italy (8):
  - Ginecologia e Fisiopatologia della Riproduzione Umana,UO Ostetricia e Ginecologia,Policlinico S.Orsola-Malpighi, Bologna
  - Ospedale Pugliese, Calabria
  - Universita degli Studi di Firenze - Azienda Ospedaliero Universitaria Careggi, DAI Materno Infantile, SOD Ginecologia e Ostetricia, Florence
  - Azienda Ospedaliero - Universitaria Policlinico di Modena, Modena
  - Universita degli Studi di Perugia - Policlinico Monteluce - Centro di Medicina Perinatale e della Riproduzione, Perugia
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Universita degli Studi di Roma La Sapienza - Umberto I Policlinico di Roma, Roma
  - Policlinico Univ. Agostino Gemelli, Roma
- Lithuania (8):
  - Saules Family Medicine Centre, Kaunas
  - UAB VAKK - Dr. Kildos Klinika, Kaunas
  - Klaipedos Miesto Poliklinika, Klaipėda
  - Public Institution Centro Poliklinika, Vilnius
  - UAB Seimos gydytojas, Vilnius
  - JSC Maxmeda, Vilnius
  - JSC Kardiolita, Vilnius
  - Vilnius University Hospital Santaros klinikos, Vilnius
- Poland (32):
  - Prywatna Klinika Polozniczo - Ginekologiczna Sp. Z O.O., Bialystok
  - Centrum Ginekologii Endokrynologii i Medycyny Rozrodu Artemida, Bialystok
  - Osrodek Badan Klinicznych IN-VIVO, Bydgoszcz
  - Przychodnia Srodmiescie Sp. z o.o., Bydgoszcz
  - Mital Site Badania Kliniczne, Elblag
  - Copernicus Podmiot Leczniczy - Szpital sw. Wojciecha, Gdansk
  - Centrum Medyczne Mikolowska Dr Adam Sipinski, Katowice
  - Clinical Medical Research sp. z o.o., Katowice
  - NZOZ Sanas, Katowice
  - Centrum Medyczne Angelius Provita, Katowice
  - Pro Familia Altera Sp. z o.o., Katowice
  - NZOZ Vita Longa Sp. z o.o., Katowice
  - Gyncentrum Sp. z o.o., Katowice
  - Pratia MCM Krakow, Krakow
  - Grazyna Bogutyn Medico Praktyka Lekarska, Krakow
  - Salve Medica-Przychodnia, Lodz
  - NZOZ Medican, Lodz
  - Centrum Medyczne Chodzki, Lublin
  - KO-MED Centra Kliniczne Sp. z o.o., Osrodek Badan Klinicznych w Lublinie II, Lublin
  - Niepubliczny Zak¿ad Opieki Zdrowotnej PROFI-MED, Lublin
  - ETYKA Osrodek Badan Klinicznych, Olsztyn
  - Centrum Innowacyjnych Terapii Sp. z o.o., Piaseczno
  - IRMED Osrodek Badan Klinicznych, Piotrkow Trybunalski
  - Clinical Research Center Spolka z ograniczona odpowiedzialnoscia Medic-R Spolka Komandytowa, Poznan
  - Estetra Study Site, Skorzewo
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin
  - Nzoz Zieniewicz Medical, Warsaw
  - Centrum Badawcze Wspolczesnej Terapii Prywatny Gabinet Lekarski Dr Anna Bochenek-Mularczyk, Warsaw
  - ETG Warszawa, Warsaw
  - Medical Concierge Centrum Medyczne, Warsaw
  - Marek Elias Gabinety Ginekologiczne, Wroclaw
  - ETG Zamosc, Zamość
- Romania (13):
  - Centrul Medical Unirea Policlinica Brasov, Brasov
  - Centrul Medical de Diagnostic si Tratament Ambulatoriu Neomed SRL, Brasov
  - SC Centrul Medical Unirea SRL, Bucharest
  - SC Quantum Medical Center SRL, Bucharest
  - Centrul Medical Euromed, Bucharest
  - Spitalul Clinic Nicolae Malaxa, Bucharest
  - Sana Monitoring, Bucharest
  - Centrul Medical Unirea - Spitalul Baneasa, Bucharest
  - Spitalul Municipal Caracal, Caracal
  - Centrul Medical Unirea, Constanța
  - Vitaplus Medclin SRL, Craiova
  - Spitalul De Urgenta Targu Mures-Emergency University County Hospital, Târgu Mureş
  - SC Centrul Medical Unirea SRL, Târgu Mureş
- Russia (11):
  - Scientific Center for Family Health Problems and Human Reproduction, Irkutsk
  - Krasnoyarsk State Medical University named after Prof. V.F. VoinoYasenetsky, Krasnoyarsk
  - LLC Olla-Med, Moscow
  - Scientific Centre Of Obsterics, Gynecology And Perinatology n.a.academican V.I.Kulakov of Federal Agency of High Tech Medical Care, Moscow
  - JCS Avicenna, Novosibirsk
  - Clinical diagnostic center Zdorovye, Rostov-on-Don
  - Saint-Petersburg State Healthcare Institution Maternity hospital, Saint Petersburg
  - The Research Institute of Obstetrics, Gynecology and Reproductology named after D.O. Ott - Center Menopause and Women's Health, Saint Petersburg
  - Astarta Clinic, Saint Petersburg
  - Woman's consulting center #22, Saint Petersburg
  - Closed Joint Stock Company Medical Company Idk, Samara
- Slovakia (2):
  - MCM GYNPED, s.r.o., Dubnica nad Váhom
  - BrenCare, s. r. o., Poprad
- Spain (4):
  - Diatros S.L.P, Gavà
  - Instituto Palacios, Salud y Medicina de la Mujer, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Virgen del Rocio, Hospital de la Mujer, Seville
- United Kingdom (11):
  - Accellacare - (MeDiNova Limited) - Northamptonshire, Corby
  - Accellacare (Previously MeDiNova) Warwickshire Quality Research Site, Coventry
  - CPS Research, Glasgow
  - Egin Research Ltd, High Wycombe
  - Queen Charlotte's and Chelsea Hospital - Imperial College Healthcare NHS Trust, London
  - Accellacare - (MeDiNova Limited) - North London, Northwood
  - Accellacare - South London, Orpington
  - Estetra Study Site, Orpington
  - Accellacare - (MeDiNova Limited) - East London, Romford
  - Accellacare - (MeDiNova Limited) - Yorkshire, Shipley
  - Accellacare - (MeDiNova Limited) - West London, Wokingham

REFERENCES:
- [Derived] Panay N, Simoncini T, Taziaux M, Bouchard C, Black A, Kapoor E, Utian W, Foidart JM, Lobo RA. Estetrol for the treatment of moderate to severe vasomotor symptoms in postmenopausal women: The design of the E4COMFORT I and II trials. Maturitas. 2026 Jan;204:108781. doi: 10.1016/j.maturitas.2025.108781. Epub 2025 Nov 17. PMID 41289787
- [Derived] Gaspard U, Taziaux M, Jost M, Coelingh Bennink HJT, Utian WH, Lobo RA, Foidart JM. A multicenter, randomized, placebo-controlled study to select the minimum effective dose of estetrol in postmenopausal participants (E4Relief): part 2-vaginal cytology, genitourinary syndrome of menopause, and health-related quality of life. Menopause. 2023 May 1;30(5):480-489. doi: 10.1097/GME.0000000000002167. Epub 2023 Feb 20. PMID 36809193